CLINICAL TRIAL: NCT02426723
Title: A Phase 1a/1b Multicenter, Open Label, Dose-Finding Study to Assess the Safety, Tolerability, Pharmacokinetics and Efficacy of CWP232291 Administered Intravenously Either Alone or in Combination With Lenalidomide and Dexamethasone in Subjects With Relapsed or Refractory Myeloma (MM)
Brief Title: Clinical Study of CWP232291 in Relapsed or Refractory Myeloma Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: JW Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JW-231MM-102
Record Dates: First submitted 2015-04-13; First posted 2015-04-27 (Estimated); Last update posted 2019-05-17 (Actual); Status verified 2019-05

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Dexamethasone

ARMS (1):
- CWP232291 (Experimental): Phase 1a: single administration of CWP232291 ,
  Phase 1b: CWP232291 combination with Lenalidomide and Dexamethasone
  Interventions: Drug: Phase 1a: CWP232291; Drug: Phase 1b: CWP232291, Lenalidomide, Dexamethasone

INTERVENTIONS:
Drug: Phase 1a: CWP232291 — CWP232291 administered alone twice weekly every 4 weeks.
Drug: Phase 1b: CWP232291, Lenalidomide, Dexamethasone — CWP232291 administered twice weekly every 4 weeks. Lenalidomide and Dexamethasone administered per standard therapy.

SUMMARY:
This is a Phase 1a/1b, multicenter, open-label, two-part study in subjects with relapsed or refractory MM:

* Phase 1a: single agent CWP232291. Dose-finding followed by cohort expansion at the maximum tolerated dose (MTD) or optimal dose as determined by the Safety Review Committee (SRC).
* Phase 1b: CWP232291 in combination with lenalidomide and dexamethasone. Dose-finding followed by cohort expansion at the combination therapy MTD or optimal dose as determined by the SRC.

ELIGIBILITY:
Inclusion Criteria:

1. Able to understand and then sign an informed consent form (ICF) prior to initiation of any study-specific procedure and treatment.
2. ≥ 18 years of age.
3. Confirmed measurable MM based on the following:

   * Serum M component (≥ 0.5 g/dL), or
   * Urine M protein ≥ 200 mg/24 hours), or
   * Serum immunoglobulin free light chains ≥ 10 mg/dL and abnormal serum immunoglobulin kappa/lambda free light chain ratio), or
   * Non-secretory disease measurable with bone marrow biopsy or radiography.
4. Failed 2 or more prior standard MM therapies, and >100 days post autologous bone marrow transplant prior to first dose for transplanted subjects. Prior lenalidomide is permitted.
5. In the absence of rapidly progressing disease, the interval from prior treatment to time of study drug administration should be ≥ 2 weeks for cytotoxic agents or at least 5 half-lives for noncytotoxic agents. Persistent clinically significant toxicities from prior chemotherapy or radiotherapy must not be greater than Grade 1.
6. Eastern Cooperative Oncology Group (ECOG) performance score 0-2 (Appendix 3).
7. Adequate bone marrow function:

   * Absolute neutrophil count (ANC) ≥ 1000/mm3, independent of growth factor support;
   * Platelet count ≥ 75,000/mm3;
   * Hb ≥ 9 g/dL (independent of transfusions or erythropoiesis-stimulating agents [ESA]).
8. Adequate renal function:

   * Serum creatinine ≤ 2.5 mg/dL;
   * Creatinine clearance (CrCl) ≥ 60 mL/minute (Cockcroft-Gault).
9. Adequate hepatic function:

   * Total bilirubin < 2.5 x upper limit of normal (ULN); direct bilirubin < 2 x ULN for Gilbert's syndrome;
   * Alkaline phosphatase (AP) ≤ 2.5 x ULN, unless considered due to organ leukemic involvement;
   * Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) ≤ 3 x ULN.

11. Women of child-bearing potential (ie, women who are premenopausal or not surgically sterile):

* Two effective forms of contraception (abstinence, intrauterine device, oral contraceptive, or double barrier device) from the time of informed consent and until at least 4 weeks after discontinuing study drugs, and
* Negative serum or urine pregnancy tests during screening and then within 3 days prior to Day 1. 12. Sexually active men - effective contraceptive methods in subject and partner from the time of informed consent and until ≥ 4 weeks after discontinuing study drugs. 13. Able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

1. Chemotherapy or immunotherapy < 5 half-lives prior to screening.
2. Not recovered to Grade 1 from adverse effects of prior myeloma therapy or radiotherapy prior to screening.
3. Systemic corticosteroids < 1 week prior to Day 1 in Phase 1a. Subjects may receive stable physiologic replacement doses of glucocorticoids (up to the equivalent of 10 mg daily prednisone) as maintenance therapy for adrenal insufficiency.
4. Uncontrolled intercurrent illness including infections and psychiatric illness/social situations that may limit compliance with protocol requirements or the evaluation of study drugs.
5. Active cardiovascular disease including myocardial infarction (MI) < 6 months of screening, symptomatic coronary artery disease (CAD), arrhythmias, hypertension, or heart failure not controlled by medication.
6. History of deep venous thrombosis and pulmonary embolism (Phase 1b).
7. Anticoagulants < 7 days prior to Day 1. Aspirin is permitted in Phase 1b per standard of care with lenalidomide-based therapy.
8. Active central nervous system (CNS) disease.
9. Known positive status for human immunodeficiency virus (HIV) and/or active hepatitis B or C.
10. Pregnant or nursing women.
11. History of hypersensitivity to lenalidomide (Part B only)
12. History of other active malignancies < 3 years prior to screening except basal cell carcinoma, low grade Gleason score ≤ 6 prostate cancer that has been removed with undetectable prostate-specific antigen (PSA), and in situ cervical carcinoma.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2015-10-19 (Actual); Primary Completion 2018-10-08 (Actual); Study Completion 2018-10-26 (Actual)

PRIMARY OUTCOMES:
Recommended dose of Phase 2 trial of CWP232291 | up to 4 weeks

SECONDARY OUTCOMES:
Cmax as a pharmacokinetic parameter of 'CWP232291' | Predose, 0.25, 0.5, 0.75, 1, 1.5 , 2 , 4 , 8, 12, 24 hours after the start of infusion
  Peak plasma concentration(Cmax) of 'CWP232291'
AUC as a pharmacokinetic parameter of 'CWP232291' | Predose, 0.25, 0.5, 0.75, 1, 1.5 , 2 , 4 , 8, 12, 24 hours after the start of infusion
  Area under the plasma concentration versus time curve (AUC) of 'CWP232291'
Cmax as a pharmacokinetic parameter of metabolites of ' CWP232204' | Predose, 0.25, 0.5, 0.75, 1, 1.5 , 2 , 4 , 8, 12, 24 hours after the start of infusion
  Peak Plasma Concentration (Cmax) of metabolites of 'CWP232291'
AUC as a pharmacokinetic parameter of metabolites of ' CWP232204' | Predose, 0.25, 0.5, 0.75, 1, 1.5 , 2 , 4 , 8, 12, 24 hours after the start of infusion
  Area under the plasma concentration versus time curve (AUC) of metabolites of 'CWP232291'

CONTACTS AND LOCATIONS:
Overall Officials: Chang-Ki Min, MD, Principal Investigator — Seoul St. Mary's Hospital; Sung-Soo Yoon, MD, Principal Investigator — Seoul National University Hospital; Jin Seok Kim, MD, Principal Investigator — Severance Hospital; Elisabet Manasanch, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (4):
- The University of Texas MD Anderson Cancer Center, Houston, Texas, United States
- South Korea (3):
  - Seoul National University Hospital, Seoul
  - Seoul St.Mary's Hospital, Seoul
  - Yonsei Severance Hospital, Seoul